CLINICAL TRIAL: NCT01627977
Title: A Descriptive Study to Evaluate the Effectiveness of the Dye Compound of the Combination of Lutein, Zeaxanthin and Brilliant Blue in Chromovitrectomy
Brief Title: Association of Lutein, Zeaxanthin and Brilliant Blue in Chromovitrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rubens Belfort Jr., Head Professor of the Departament of Ophthalmology, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LUT-RET
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Epiretinal Membrane; Macular Hole; Proliferative Diabetic Retinopathy
Keywords: chromovitrectomy; epiretinal membrane
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations | interventions — Zeaxanthins; brilliant blue; Lutein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dye of Lutein/Zeaxanthin/Brilliant Blue (Experimental): during the surgery will be evaluated if the dye is suitable for dyeing the internal limiting membrane as well as the epiretinal membrane
  Interventions: Other: Dye of Lutein, Zeaxanthin and Brilliant Blue

INTERVENTIONS:
Other: Dye of Lutein, Zeaxanthin and Brilliant Blue — dye composed of Lutein, Zeaxanthin and Brilliant Blue will be used during the vitrectomy surgery to dye the membranes
  Other Names: lutein, zeaxanthin, brilliant blue

SUMMARY:
The aim of this study is to test the efficacy of the combination of dye Lutein, Zeaxanthin and brilliant blue to stain the internal limiting membrane as well as the epiretinal membranes during the Vitrectomy surgery.

DETAILED DESCRIPTION:
Twenty five patients with epiretinal membrane, macular hole or proliferative diabetic retinopathy and indication of vitrectomy surgery will be selected to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, both gender
* Diagnosis of epiretinal membrane OR macular hole OR proliferative diabetic retinopathy
* Indication of surgical treatment for removal of the epiretinal membrane

Exclusion Criteria:

* Any history of eye disease
* glaucoma
* Eye infection affecting any structure provided eye

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Visibility of the membrane after injection of the dye | during the surgery
  The visibility of the membrane after injection of the dye should be graduated by the physician as Bad, OR Fair, OR Good, OR Very Good

SECONDARY OUTCOMES:
Degree of impregnation of the dye | during the surgery
  The degree of impregnation of the membrane by the dye should be graduated according to the following scale:(0)not flushed; (1)stained weakly (light green); (2)moderately stained (medium green); (3)stained intensely (dark green)
Usefulness of the dye | at the end of surgery
  the physician should evaluate the usefulness of the dye, according to the following scale: Bad, Fair, Good, Very Good

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Depto. of Ophthalmology - Hospital São Paulo - UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
data published: Graefes Arch Clin Exp Ophthalmol. 2014 Jul;252(7):1071-8.

REFERENCES:
- [Derived] Badaro E, Furlani B, Prazeres J, Maia M, Lima AA, Souza-Martins D, Muccioli C, Lucatto LF, Belfort R Jr. Soluble lutein in combination with brilliant blue as a new dye for chromovitrectomy. Graefes Arch Clin Exp Ophthalmol. 2014 Jul;252(7):1071-8. doi: 10.1007/s00417-013-2539-5. Epub 2014 Jan 19. PMID 24441951